CLINICAL TRIAL: NCT02089932
Title: The Effects of Different Dose Levels of Peri-neural Dexmedetomidine on the Pharmacodynamic and Side Effects Profiles of Bupivacaine-induced Ultrasound-guided Femoral Nerve Block
Brief Title: Dexmedetomidine in Different Dose Levels as Adjuvant to Bupivacaine-induced Ultrasound-guided Femoral Nerve Block.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Nassar,MD, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N-60-2013
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Dexmedetomidine; Femoral Nerve Block; Arthroscopic Knee Surgery
Keywords: femoral nerve block; peri-neural dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group B: control bupivacaine group (Placebo Comparator): Patient in this group will receive 25 ml bupivacaine 0.5% plus 1 ml normal saline peri-neurally
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block; Drug: Placebo
- Group B-DEX 25 : Peri-neural Dexmedetomidine (Experimental): Patients in this group will receive 25 ml of 0.5% bupivacaine plus 1 ml (25 microgram) Dexmedetomidine peri-neurally
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block
- Group B-DEX 50:Peri-neural Dexmedetomidine (Experimental): Patients in this group will receive 25 ml of 0.5% bupivacaine plus 1 ml (50 microgram) Dexmedetomidine peri-neurally
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block
- Group B-DEX 75:Peri-neural Dexmedetomidine (Experimental): Patients in this group will receive 25 ml of 0.5% bupivacaine plus 1 ml (75microgram) Dexmedetomidine peri-neurally
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block

INTERVENTIONS:
Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block — ultrasound guided femoral nerve block with injection of 25 ml bupivacaine 0.5% perineurally with 1 ml dexmedetomidine 25, 50, or 75 microgram perineurally.
  After adequate assessment of femoral nerve block, patients will be transferred to the operating room to receive a standard general anesthesia.
Drug: Placebo
  Arms: group B: control bupivacaine group

SUMMARY:
The duration of sensory block after single dose of long acting local anesthetics is not sufficient to avoid the postoperative use of opioids. Alpha-2 adrenoceptor agonists such as clonidine have been shown to increase the duration of peripheral nerve block. Dexmedetomidine is a more potent and selective α-2-adrenoceptor compared to clonidine. To the best of our knowledge, the use of Dexmedetomidine in different dose levels as adjuvant to local anesthetic was not previously reported for femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

* all patients with ASA physical status I or II, scheduled for arthroscopic knee surgery

Exclusion Criteria:

* Patients who are refusing regional block, patients with diabetic peripheral neuropathy, renal or hepatic dysfunction, inflammation or infection at the puncture site, and history of allergic reaction to study medications

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
duration of sensory block | Every 5 minutes for the first 30 minutes after end of study medications injection, then postoperatively every 2 hours till complete recovery of normal sensation.
  the time interval between the onset of the sensory block and the complete resolution of normal sensation. Over a period of 30 min after injection of the study medications and every 2 hours postoperatively till complete recovery of normal sensation; a blinded investigator will assess sensory block with pinprick test using a 3-point scale: 0 ═ complete loss of sensation, 1 ═ partial loss of sensation and 2 ═ normal sensation. Pinprick test will be done in comparison to the contralateral area at the sensory distribution of the femoral nerve.

SECONDARY OUTCOMES:
Time to first request of postoperative rescue analgesic | over the first postoperative 24hours
  the time interval between the onset of successful sensory block and the first request to postoperative analgesia
Onset of sensory block | up to 30 minutes after the end of injection
  the time elapsed between the end of injection and the development of complete sensory block
Onset of motor block | up to 30 minutes after the end of injection
  the time elapsed between the end of injection and the development of complete motor block
visual analogue pain scores (VAS) | 2hours post operative and for 24hours
  Visual analogue pain scores (resting and dynamic VAS) will be assessed at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively.
Richmond Agitation-Sedation Score (RASS) | 2hours post operative and for 24hours
  Richmond Agitation-Sedation Score (RASS) will be assessed at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively.
duration of motor block | Every 5 minutes for the first 30 minutes after end of study medications injection, then postoperatively every 2 hours till complete recovery of motor power.
  The time interval between the onset of the motor block and the complete resolution of the motor power in quadriceps muscle. Over a period of 30 min after injection of the study medications and every 2 hours postoperatively till complete recovery of motor power; a blinded investigator will assess the motor block using a 3-point scale where: 0 ═ no movement, 1 ═ reduced motor strength, but some perceptible movement, and 2 ═ normal motor function.
total morphine consumption | The first 24 hours postoperatively
  The total dose of morphine needed by the patient postoperatively till 24 hours.
perioperative hemodynamic parameters | will be recorded at 0, 15, 30 minutes after femoral nerve block, then every 10 minutes intraoperatively, and every 2 hours postoperative for a period of 12 hours.
  Vital signs (heart rate and arterial blood pressure) will be recorded at 0, 15, 30 minutes after femoral nerve block, then every 10 minutes intraoperatively, and every 2 hours postoperative for a period of 12 hours.
incidence of side effects. | from the injection time till 24 hours postoperatively
  Adverse events will be defined as hypotension (a 30% decrease in systolic blood pressure in relation to the baseline value), bradycardia (heart rate less than 60 beats per minute), desaturation (SpO2 < 90% on room air) and postoperative nausea and/or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, Professor of Anesthesia, Study Chair — Cairo University
Locations (1):
- Kasr Al Ainy, Cairo, Egypt